CLINICAL TRIAL: NCT01848626
Title: Study With Advanced Vaginal Tactile Imager
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: VTI 04
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Investigative Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are:

1. To collect data necessary for assessing the performance of advanced Vaginal Tactile Imager (VTI) and evaluating the probe ergonomic design, safety and patient tolerance;
2. To assess the clinical suitability of the interface software to facilitate the data collection process and to get in vivo examination data for validation of visualization and analysis routines;
3. To test the data collection technique and establish a reliable examination procedure.

ELIGIBILITY:
Inclusion Criteria:

Adult women (over the age of 21) falling within one of the following groups:

1. No evidence of pelvic floor disorder and no prior pelvic surgery;
2. Stage 1 or 2 pelvic organ prolapse affecting one or more vaginal compartment.

Exclusion Criteria:

1. Active skin infection or ulceration within the vagina
2. Presence of a vaginal septum;
3. Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder;
4. Ongoing radiation therapy for pelvic cancer;
5. Impacted stool;
6. Recent (less than three months) pelvic surgery;
7. Significant pre-existing pelvic pain including levator ani syndrome, severe vaginismus or vulvodynia;
8. Severe hemorrhoids;
9. Surgically absent rectum or bladder;
10. Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult females, presenting to the urogynecological office for a vaginal examination with normal pelvic floor organs, referred to gynecologic examination due to pelvic organ prolapse concern or earlier diagnosed with pelvic organ prolapse, will be considered eligible as volunteers to be enrolled in the clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Imaging performance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, PhD, Principal Investigator — Artann Laboratories
Locations (1):
- Princeton Urogynecology, Princeton, New Jersey, United States

REFERENCES:
- [Derived] van Raalte H, Egorov V. Characterizing female pelvic floor conditions by tactile imaging. Int Urogynecol J. 2015 Apr;26(4):607-9. doi: 10.1007/s00192-014-2549-9. Epub 2014 Oct 25. PMID 25344223